CLINICAL TRIAL: NCT00851578
Title: ASA Plavix Feasibility Study With WATCHMAN Left Atrial Appendage Closure Technology
Acronym: ASAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ST1056
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2013-09

CONDITIONS: Atrial Fibrillation
Keywords: AF; atrial fibrillation; LAA occlusion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WATCHMAN (Experimental): non-valvular atrial fibrillation patients contraindicated to warfarin
  Interventions: Device: WATCHMAN

INTERVENTIONS:
Device: WATCHMAN — WATCHMAN LAA Closure Device

SUMMARY:
The purpose of the study is to characterize the performance of the WATCHMAN LAA Closure Device in atrial fibrillation patients for which long term warfarin therapy is contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* paroxysma, persistent, or permanent non-vlavular atrial fibrillation
* contraindicated to warfarin
* eligible for clopidogrel, ticlopdine, heparin, or aspirin
* CHADS score 1 or greater

Exclusion Criteria:

* NYHA Class IV
* LAA obliteration
* Heart transplant
* LVEF less than 30%
* greater than 50% carotid stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Feasibility study to characterize the performance of the WATCHMAN LAA Closure device in atrial fibrillation patients contracindicated to warfarin treatment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- NA Homolce Hospital, Prague, Czechia
- Germany (3):
  - Sankt Katharinen Hospital / Cardiovasculares Centrum, Frankfurt
  - Herzzentrum Leipzig, Leipzig
  - Chefarzt der Medizinischen Klinik III/Kardiologie, Regensburg

REFERENCES:
- [Derived] Reddy VY, Mobius-Winkler S, Miller MA, Neuzil P, Schuler G, Wiebe J, Sick P, Sievert H. Left atrial appendage closure with the Watchman device in patients with a contraindication for oral anticoagulation: the ASAP study (ASA Plavix Feasibility Study With Watchman Left Atrial Appendage Closure Technology). J Am Coll Cardiol. 2013 Jun 25;61(25):2551-6. doi: 10.1016/j.jacc.2013.03.035. Epub 2013 Apr 10. PMID 23583249